CLINICAL TRIAL: NCT05982808
Title: A Novel Surgical Technique of CLIF Correction VS. Conventional Corrective Strategy on the Treatment of Adult Complex Spinal Deformity With a Multicenter Randomized Controlled Trial
Brief Title: CLIF Correction VS. Conventional Correction Strategy for ASD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Wang Zhiwei, MD, Principal Investigator, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIF correction for ASD
Record Dates: First submitted 2023-07-31; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Spinal Deformity
Keywords: adult spinal deformity; CLIF; crenal lumbar interbody fusion; minimal invasive; correction; surgical strategy

STUDY DESIGN:
Intervention Model Description: with/without novel CLIF correction
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel CLIF correction (Experimental): ASD patients with novel CLIF correction
  Interventions: Procedure: CLIF correction
- conventional correction strategy (Active Comparator): ASD patients with conventional correction strategy
  Interventions: Procedure: conventional correction strategy

INTERVENTIONS:
Procedure: CLIF correction — CLIF correction was a novel surgical techqiue of correction of spinal deformtiy with minimal invasive approach
  Arms: Novel CLIF correction
Procedure: conventional correction strategy — conventional correction was the classic surgical techqiue of correction of spinal deformtiy with open posterior approach
  Arms: conventional correction strategy

SUMMARY:
The present study intends to: 1）establish a multi-center large-sample randomized controlled trial to explore the technical advantages and surgical indications of the novel surgical technique of CLIF correction for ASD compared with the conventional correction strategy; 2）analyze the postoperative clinical and imaging results, and to explore the related complications and preventive measures; 3） establish 2-year follow-up to further quantify the clinical and radiographical outcomes of CLIF correction.

DETAILED DESCRIPTION:
Adult spinal deformity (ASD) is the most common spinal deformity in the elder, which often causes the low back pain and/or physical deformity. Severe cases need surgical treatment. Because the conventional posterior approach had the disadvantages of big trauma and slow recovery, and the elder were always complicated with complicated medical diseases, the perioperative risk was high. At present, the novel surgical technique of CLIF correction was a popular way for ASD treatment. Preliminary results showed that it had less trauma, shorter operation time, faster recovery, fewer complications and remarkable clinical and adiographical outcomes. Therefore, the present study intends to: 1) establish a multi-center large-sample randomized controlled trial to explore the technical advantages and surgical indications of the novel CLIF correction for ASD treatment compared with the conventional correction strategy; 2) establish 2-year follow-up to further quantify the clinical and radiographical outcomes, and to explore the related complications and preventive measures;. Therefore, the present project aims to explore the best surgical plan for treating ASD by studying the safety and effectiveness of the novel CLIF correction, and provide new surgical strategies for minimally invasive and Individualized treatment for ASD.

ELIGIBILITY:
Inclusion Criteria:

* adult spinal deformtiy;
* 40yrs≤age≤80yrs;
* Lenke-Silva classification II-V grade;
* ineffective with conservative treatment;

Exclusion Criteria:

* severe osteoprosis with T value <-2.5;
* with preliminary spinal surgery;
* ASA score≥III grade;
* more than II degree spondylisthesis;
* with mental disease;

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
ODI score | 2 year after surgery
  ODI score is Oswestry Disability Index（0-100）, indicating the back pain; the higher score, the greater back pain

SECONDARY OUTCOMES:
SF-36 score | 2 year after surgery
  SF-36 score is the MOS item short from health survey (0-100), indicating the life quality; the higher score, the better life quality

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-wei WANG, Ph.D and MD., Principal Investigator — 2nd Hospital, Zhejiang University, School of Medicine
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
When the first stage is done, the study plan would be open for others

REFERENCES:
- [Result] Aebi M. The adult scoliosis. Eur Spine J. 2005 Dec;14(10):925-48. doi: 10.1007/s00586-005-1053-9. Epub 2005 Nov 18. PMID 16328223
- [Result] Ailon T, Smith JS, Shaffrey CI, Lenke LG, Brodke D, Harrop JS, Fehlings M, Ames CP. Degenerative Spinal Deformity. Neurosurgery. 2015 Oct;77 Suppl 4:S75-91. doi: 10.1227/NEU.0000000000000938. PMID 26378361
- [Result] Schwab F, Dubey A, Gamez L, El Fegoun AB, Hwang K, Pagala M, Farcy JP. Adult scoliosis: prevalence, SF-36, and nutritional parameters in an elderly volunteer population. Spine (Phila Pa 1976). 2005 May 1;30(9):1082-5. doi: 10.1097/01.brs.0000160842.43482.cd. PMID 15864163
- [Result] Smith JS, Shaffrey CI, Glassman SD, Berven SH, Schwab FJ, Hamill CL, Horton WC, Ondra SL, Sansur CA, Bridwell KH; Spinal Deformity Study Group. Risk-benefit assessment of surgery for adult scoliosis: an analysis based on patient age. Spine (Phila Pa 1976). 2011 May 1;36(10):817-24. doi: 10.1097/BRS.0b013e3181e21783. PMID 20683385